CLINICAL TRIAL: NCT05226715
Title: Immediate Effect of Lower Extremity Joint Manipulation on a Lower Extremity Somatosensory Illusion: a Preliminary, Randomized, Controlled Crossover Clinical Trial
Brief Title: Effect of Lower Extremity Joint Manipulation on a Lower Extremity Somatosensory Illusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parker University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Parker
Record Dates: First submitted 2021-11-01; First posted 2022-02-07 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Coordination and Balance Disturbances; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Received a bilateral, lower extremity manipulation series
  Interventions: Other: chiropractic manual therapy
- Control (No Intervention): 30 seconds of lying supine on a chiropractic bench (control) without manual manipulation

INTERVENTIONS:
Other: chiropractic manual therapy — high velocity low amplitude thrust into a human joint
  Arms: Intervention

SUMMARY:
The purpose of this study is to examine the influence of extremity manipulation on individual's center of pressure after they adapt to an ankle based illusion.

ELIGIBILITY:
Inclusion Criteria:

* No previous surgeries
* Not knowingly pregnant
* No neuromusculoskeletal injuries or systemic diseases that could affect an individual's ability to stand on an incline for 3 minutes with their eyes closed.

Exclusion Criteria:

- Weight over the force plate operating limit of 440 lbs

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-05-16 (Actual); Study Completion 2021-05-16 (Actual)

PRIMARY OUTCOMES:
Center of pressure position | baseline, immediately post-intervention, same day
  position in centimeters as evaluated by a force plate

SECONDARY OUTCOMES:
Pathlength | baseline, immediately post-intervention, same day
  cumulative distance traveled by center of pressure during trial
RMS | baseline, immediately post-intervention, same day
  (Root mean square) measure of amplitude of center of pressure during trial
Mean velocity | baseline, immediately post-intervention, same day
  average speed and direction of center of pressure during trial

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Malaya, DC, Principal Investigator — Parker University
Locations (1):
- Synapse Laboratory, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schueren S, Hunger H, Pham H, Smith DL, Layne C, Malaya CA. Immediate effect of lower extremity joint manipulation on a lower extremity somatosensory illusion: a randomized, controlled crossover clinical pilot study. Front Hum Neurosci. 2022 Nov 8;16:1011997. doi: 10.3389/fnhum.2022.1011997. eCollection 2022. PMID 36425882